CLINICAL TRIAL: NCT04442438
Title: Moral Case Deliberation on the Intensive Care: Effect of Implementation of a Moral Case Delibration Meetings on the Prevalence of Burn-out Syndrome in the ICU
Brief Title: Effect of Implementation of a Moral Case Delibration Meetings on the Prevalence of Burn-out Syndrome in the ICU
Acronym: MCDIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Marieke Zegers, Principal Investigator, Radboud University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CH2018-01
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Burnout, Professional; Caregiver Exhaustion
Keywords: Moral case deliberation; Moral distress; Cohort study; Intensive care units; Quality of care; Moral development; Organizational culture
MeSH Terms: conditions — Burnout, Professional; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Longitudinal Stepped Wedge cluster randomized Trial with an open cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Intensive care unit 1 (Experimental): Receives of intervention consisting of monthly moral case deliberation (ethical decision-making) meetings, planned and set up by ICU professionals which have received the task of being more attentive to ethical situations during work.
  Interventions: Other: Monthly moral case deliberation
- Intensive care unit 2 (Other): First non-intervention, then flips to experimental arm type after six months.
  Interventions: Other: Monthly moral case deliberation
- Intensive care unit 3 (Other): First non-intervention, then flips to experimental arm type after six months.
  Interventions: Other: Monthly moral case deliberation
- Intensive care unit 4 (Other): First non-intervention, then flips to experimental arm type after twelve months.
  Interventions: Other: Monthly moral case deliberation
- Intensive care unit 5 (Other): First non-intervention, then flips to experimental arm type after twelve months.
  Interventions: Other: Monthly moral case deliberation
- Intensive care unit 6 (Other): First non-intervention, then flips to experimental arm type after Eighteen months.
  Interventions: Other: Monthly moral case deliberation

INTERVENTIONS:
Other: Monthly moral case deliberation — Once per month, ICU professionals will take part in moral case deliberation. As part of the intervention, two or three ICU professionals (physicians and nurses) are tasked with selecting a case for moral discussion. Moral case deliberation is attended by around thirty individuals per month per unit. A feedback system will be developed used to spread the knowledge/insights from the case deliberation to all professionals in the unit.

SUMMARY:
Burnout syndrome (BOS) has a high prevalence in critical care nurses and physicians. Both personal characteristics and work-related factors have been associated with BOS. Despite this high prevalence of burnout and its potential for serious consequences, few studies have tested interventions to address the problem. Whereas person-directed interventions may be effective for periods less than 6 months, changes in the organization tend to have a longer lasting effect. Lack of participation in morally complex decision-making is assumed to be an important risk factor for the development of burnout symptoms. Implementation of structured, multi-professional medical ethical decision-making - so called moral case deliberation (MCD) - is proven feasible in an ICU setting. Health care workers involved in patient care perceived that active participation in ethical decision making resulted in better awareness of the background of the individual decisions and improved understanding of the ethical dilemma. The effects of this intervention on health-care workers well-being was not investigated.

DETAILED DESCRIPTION:
Studies have shown that healthcare professionals working at the ICU are exposed to greater risk of developing burnout than colleagues working in other fields of medicine (Moss, Good, Gozal, Kleinpell, & Sessler, 2016). It is widely suggested that moral distress, resulting from morally problematic situations particular for the ICU, is an important risk factor for burnout (Fumis, Junqueira Amarante, de Fatima Nascimento, & Vieira Junior, 2017). One suggested way to help caregivers mitigate moral distress is moral case deliberation. Moral case deliberation is a structured dialogue between healthcare providers about ethically problematic situations in their daily practice. It has been widely held that frequent moral case deliberation may help healthcare providers to better appreciate moral problems, to learn about their own and others' moral viewpoints, to foster a sense cohesion within their team and to mitigate moral distress (Haan, van Gurp, Naber, & Groenewoud, 2018). Moral case deliberation may particularly help professionals if it is based on professionals' own objectives in and experiences and expectations of moral case deliberation. It is therefore needed to firmly root moral case deliberation in the ICU practice together with/with the help of ICU-professionals (Weidema, van Dartel, & Molewijk, 2016). Healthcare professionals themselves are best able to evaluate, learn from and adjust the practice of moral case deliberation on the ICU.

This research sets out to assess the claim that moral case deliberation can help mitigate moral distress among healthcare providers and as such reduce the risk of burnout. It does so by employing Mixed Methods Action Research (MMAR), through which the research will be conducted through and with ICU-professionals, creating co-ownership of moral case deliberation among participants. The study hopes to achieve that, instead of developing burnout as a consequence of moral distress, moral case deliberation will help IC professionals learn from morally distressing situations, potentially leading to cultural an organizational improvement and improvement of quality of care.

Research questions to be answered:

1. How does moral distress, as a supposed risk factor for burnout of IC-professionals, relate to other risk factors of burnout, personality, negative work-home interactions and the ICU context?
2. How do IC-professionals experience preparation, participation and the impact on daily practice of particular moral case deliberations?
3. Does moral case deliberation lead to a reduction of moral distress, burnout and team cohesion?
4. How can IC-professionals establish cumulative learning from moral case deliberation throughout their department?

Methods:

Quantitative methods Quantitative methods will be used to assess questions 1 and 3. Survey data will be gathered in a stepped wedge trial. Surveys will be sent to around 450 ICU-professionals which are nested in six ICUs, nested in two hospitals. The data thus has a multilevel structure (individuals in units in hospitals). The study aims for a response rate of 50% or higher, including more than 230 participants. This is expectation is formulated on the basis of the departments' experience of response rates in previous studies done in this population. During the trial, the different ICUs will receive the intervention in a stepwise manner. Within a stepped wedge design, what is randomized is the time point at which a unit receives the intervention. One unit starts in January 2020 and will receive the intervention for the full two years. Two units will start participating as of July 2020 and will then participate until December 2021. In January 2021, two other units will start participating. The last unit will receive the intervention as of July 2021 and participate for the remaining six months.

Survey data will be gathered at five measurement points, after every 6 months, the first being a baseline measurement. The baseline measurement will take place before January 2020, the second measurement will take place before July 2020, the third measurement will take in the months preceding January 2021, the fourth measurement will take place in the months preceding July 2021 and the last measurement will take place in December 2021. The survey consists of validated measurements for burnout syndrome (UBOS-C), moral distress (MDS-R), work-home interaction (SWING), personality (BFI), departmental culture (Culture of Care Barometer) and team cohesion (a set of six questions taken from the Safety Attitudes Questionnaire).

The baseline data will inspire answering research question 1. Hierarchical linear regression analysis will be used to assess the association between several concepts (e.g. moral distress, work-home interaction, personality). With hierarchical regression analysis, the explaining variance of moral distress on burn-out, controlled for burnout risk factors such as work-home interaction and personality, will be analysed. Hierarchical linear regression is a framework for model comparison: several regression models are built by adding variables to previous model at each new step and thus, later models always include the previous smaller models. The question is whether the newly added variable shows a significant improvement in the proportion of explained variance of burnout (the R2).

The survey data gathered at all five measurement points is suited for analysis which allows for assessment of question 3. The data gathered in the stepped wedge design, in which clusters (units) are randomized, is well suited for interrupted time series analysis. Interrupted time series analysis is used to evaluate the effect of an intervention in longitudinal data. The key assumption of interrupted time series analysis of this data is that moral case deliberation, as an intervention, changes the pre-intervention trend of burnout prevalence among ICU-professionals; in other words, it assumes that the pre-intervention trend would continue unchanged into the post-intervention period if there had not been an intervention. Training, as well as the advice of an expert statistician (Steven Teerenstra), will be sought to gain better insight in conducting interrupted time series analysis.

ELIGIBILITY:
Inclusion Criteria:

* ICU professionals age 16 years or older working in intensive care departments in the Radboud University Medical Centre or the Canisius Wilhelmina Hospital
* gave written informed consent

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Burnout - measured by the Utrecht Burnout Scale (UBOS-C) survey instrument | six months
  An excessive reaction to stress caused by one's environment that may be Burnout is characterized by feelings of emotional and physical exhaustion, coupled with a sense of frustration and failure. This is measured through the Utrecht Burnout Scale (UBOS-C) survey instrument, a Dutch version of the Maslach Burnout Inventory (MBI), containing 20 items. The MBI measures three dimensions of burnout: emotional exhaustion, depersonalisation and personal accomplishment on 0 to 6 scales. Higher scores on emotional exhaustion and depersonalisation mean a worse outcome, while a higher score on personal accomplishment means a better outcome.

SECONDARY OUTCOMES:
Moral distress - measured by the 21-item moral distress scale (revised version) survey instrument | six months
  Moral distress is the emotional state that arises from a situation when an ICU professional feels that the ethically correct action to take is different from what he or she is tasked with doing. When policies or procedures prevent a professional from doing what he or she thinks is right, that presents a moral dilemma. Moral distress will be measured by the moral distress scale, a survey instrument containing 21 items. Participants are asked to rate all these situations in terms of frequency and intensity on scales ranging from 0 to 4. A total moral distress scale is calculated by multiplying frequency and intensity and adding all items together, which makes up a score between 0 and 336. A higher value means a worse outcome.

OTHER OUTCOMES:
Team cohesion - measured by the Team Climate Inventory survey instrument | six months
  Degree to which participants feel that they are part of a team. It is measured throuhg the Team Climate Inventory survey instrument, a survey instrument containing 6 items.

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Van Gurp, PhD, Principal Investigator — IQ healthcare, Radboud University medical center; Hans Van der Hoeven, MD, PhD, Principal Investigator — Intensive care, Radboud Univesity medical center
Locations (2):
- Netherlands (2):
  - Radboud university medical centre, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kok N, Zegers M, Teerenstra S, Fuchs M, van der Hoeven JG, van Gurp JLP, Hoedemaekers CWE. Effect of Structural Moral Case Deliberation on Burnout Symptoms, Moral Distress, and Team Climate in ICU Professionals: A Parallel Cluster Randomized Trial. Crit Care Med. 2023 Oct 1;51(10):1294-1305. doi: 10.1097/CCM.0000000000005940. Epub 2023 Jun 5. PMID 37272981